CLINICAL TRIAL: NCT05506345
Title: Research on the Application Effect of Creative Drama Workshop Based on Social Interaction Theory in Clinical Practice Nursing Students' Stress Management
Brief Title: Research on the Effect of Drama Workshop on Stress Management of Nursing Students Based on Social Interaction Theory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiaxing Zhou (Other)
Responsible Party: Sponsor-Investigator, Jiaxing Zhou, Bachelor of Science in Nursing, Affiliated Hospital of Jiaxing University
Organization: Affiliated Hospital of Jiaxing University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FirstHJiaxing
Record Dates: First submitted 2022-08-14; First posted 2022-08-18 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The intervention group carried out a series of creative drama workshops based on social interaction theory on the basis of routine nursing teaching.
  Interventions: Behavioral: Creative Drama Workshop
- control group (No Intervention): The control group adopted conventional nursing teaching methods (conventional nursing teaching methods included safety education, healthy lifestyle, role positioning of nursing students, nursing etiquette, communication skills, nursing professional theory and skill training, nursing career planning, and clinical one-on-one teaching, according to plan to complete the teaching task).

INTERVENTIONS:
Behavioral: Creative Drama Workshop — * The host introduces the theme and stressor scene of this workshop
    * Nursing students group discussion
      * Nursing student group performance practice ④Nursing group formal performance ⑤Nursing student group discussion ⑥The representative of the nursing student group made a speech ⑦ The host summarizes the positive coping methods of nursing students in stressor events
  Arms: intervention group

SUMMARY:
Background: Nursing interns are the backup force for the development of the nursing career and the main force of the future nursing team. Different pressures will arise due to changes in the environment, schedule and interpersonal relationships. Stress will negatively affect nursing students, leading to anxiety, depression and even despair, which will accelerate the brain drain and shortage in the nursing industry, and is extremely detrimental to the healthy development of the nursing workforce.

Objective: To explore the effect of creative drama workshop on the stress level and stress coping behavior of nursing students.

Methods: The intern nursing students who met the standards were randomly divided into an intervention group and a control group. Both groups received routine nursing training, and the intervention group participated in creative drama workshops on this basis. The stress levels and stress coping styles of the two groups of nursing students were evaluated before and after the intervention and once a month during the intervention using the Nursing Student Stressor Scale and the Simple Coping Style Scale.

DETAILED DESCRIPTION:
At present, the research on nursing student stress at home and abroad mainly focuses on the source of stress and the adverse consequences of excessive stress on nursing students. At first,stressors mainly come from a negative social environment; poor psychological resilience; heavy work tasks and caring for patients suffering from physical and mental illness; low interest in clinical practice; employment pressure; adverse nursing events; hospital violence. In addition, studies have shown that the degree of death anxiety among trainee nursing students is higher than that of general medical students, and they have different degrees of death anxiety and psychological fluctuations when the patient dies. Then the impact of stress on nursing students: Stress has a negative impact on nursing students' professional identity; academic and internship performance, sleep and quality of life, and physical and mental health, and may even affect their future careers in the nursing industry. Research by Zeng Xiaofeng and Alshawush has shown Excessive stress can increase nursing students' willingness to leave. With the growing age of baby boomers and the growing demand for medical care, the nursing industry is already facing a shortage of human resources. It is very unfavorable to the construction of the nursing team and the healthy development of the industry.

The stress management for nursing students has been explored and practiced at home and abroad. Domestic researches are basically limited to the psychological decompression of nursing students in specific specialized disciplines or in specific situations. Some studies have used situational simulation teaching to reduce the occurrence of negative psychological states and work adjustment disorders of nursing students, and help students prepare psychologically for work pressure. Although some studies are aimed at the whole group of nursing students during the internship period, the intervention time is short and is not combined with stressors. For example, Yan Yuzhu's team discussed the effect of peer support groups on relieving the pressure of intern nursing students, and it played a certain role in relieving the pressure of intern nursing students, but the intervention time was only 3 months, and the intervention period was relatively short. However, changing established behaviors is a complex process, and the impact of interventions on internship nursing students should be a continuous process, and any stress management intervention should reflect the continuity of the process. Relatively speaking, there are many foreign intervention studies on the stress of interns. For example, Noh GO and others study the effect of SBAR (situation, background, assessment and recommendation) and the combination of SBAR and self-confidence training, reducing clinical practice stress by improving communication skills; Yuksel A's team and Lu J F's team used mindfulness interventions to reduce nursing students' stress levels; in addition, progressive muscle relaxation training was shown to improve the psychosocial responses to nursing student stress and burnout, but these were all aimed at reducing stress, Interventional research on reducing the stress level of nursing students has not focused on how to improve the self-stress management ability and stress coping behavior of nursing students.

Forum theatre, as a teaching form of applied drama, uses it to manage the conflict situations encountered by nursing students in clinical practice, and has received good feedback from nursing students. Through forum games, the conflict situations encountered by trainee nursing students during clinical practice can be narrated and explored in a powerful way, providing a good opportunity to further improve the quality of nursing education . Forum theatre has been successfully applied internationally in educational subjects in different fields, with good results in healthcare education for nursing, midwifery and medical students . In conclusion, drama is a powerful educational tool with unique advantages, and the application of its science to stress management in nursing interns is worth exploring.

This study intends to construct a creative drama workshop program based on social interaction theory, and to explore its role in improving the stress coping ability of nursing students and reducing the stress level of nursing students through the implementation of the program. This method is used to explore its effect on the stress management of clinical practice nursing students, so as to reduce their stress level, improve their stress coping style, and improve their management level of stress, so that they can obtain a positive work experience and prevent the stress of nursing students in a targeted manner. High stress that negatively affects occupational mood and work ability, and preventing other adverse effects caused by excessive stress, is of great significance to the development of nursing students and the nursing profession.

ELIGIBILITY:
Inclusion Criteria:

Participate in this study voluntarily and sign the informed consent Nursing students in full-time college and undergraduate clinical practice period Clear thinking and normal comprehension ability

Exclusion Criteria:

Withdrawal from the researcher for other reasons Those with previous mental illness or mental illness during the internship.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Nursing student stress level | 8 months
  The Nursing Student Stressors Scale prepared by Zhang Guixia et al. was used, and a Likert 5-point scale was used, with 1 to 5 points indicating the degree of stress caused by the survey items to the nursing students, ranging from weak to strong. The reliability of the scale is Cronbach's alpha of 0.820, and the test-retest reliability r is 0.823; it has good construct validity.
stress coping style | 8 months
  The simple coping style questionnaire prepared by Xie Yaning adopts self-assessment method, adopts Likert 4-level scoring method, does not use, occasionally uses, sometimes uses and often uses (respectively 0, 1, 2, 3 points), Higher scores indicate more frequent adoption. The scale Cronbach's coefficient a=0.90, of which the positive coping subscale a=0.89, the negative coping subscale a=0.78, and the test-retest reliability is 0.89, which has high reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jiaxing (Affiliated Hospital of Jiaxing University), Jiaxing, Zhejiang, China